CLINICAL TRIAL: NCT02777320
Title: Comparison of Intravenous Ibuprofen and Paracetamol in Patients With Sciatica Presented to the Emergency Department: A Randomized, Double-Blind, Controlled Trial.
Brief Title: Comparison of Intravenous Ibuprofen and Paracetamol in Patients With Sciatica Presented to the Emergency Department
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Mustafa Serinken, professor, Pamukkale University
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: Sciatica-IvsP
Record Dates: First submitted 2016-05-17; First posted 2016-05-19 (Estimated); Last update posted 2016-07-15 (Estimated); Status verified 2016-07

CONDITIONS: Sciatica
Keywords: Sciatica; Ibuprofen; Paracetamol; Emergency Medicine
MeSH Terms: conditions — Sciatica | interventions — Acetaminophen; Ibuprofen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- paracetamol group (Experimental): First Group: 1000 mg Paracetamol in 150 ml normal saline given as a slow intravenous infusion over 5 minutes. (100 ml of saline is removed before the addition of the 100 ml paracetamol to be the same volume)
  Interventions: Drug: paracetamol
- Ibuprofen group (Experimental): Second Group: 400 mg Ibuprofen in 150 ml normal saline given as a slow intravenous infusion over 5 minutes
  Interventions: Drug: Ibuprofen

INTERVENTIONS:
Drug: paracetamol — 1000 mg Paracetamol in 150 ml normal saline given as a slow intravenous infusion over 5 minutes (100 ml of saline is removed before the addition of the 100 ml paracetamol to be the same volume)
  Other Names: Perfalgan; Partemol; Parol
  Arms: paracetamol group
Drug: Ibuprofen — 400 mg Ibuprofen in 150 ml normal saline given as a slow intravenous infusion over 5 minutes
  Other Names: Intrafen; Caldolon
  Arms: Ibuprofen group

SUMMARY:
Currently, Paracetamol and Ibuprofen are widely used by emergency physicians in Turkey for the pain treatments.

The objective of the study was to assess whether intravenous Paracetamol has superior Sciatica pain reduction will compare with Ibuprofen in emergency department (ED) adults.

Half of the participants will receive Paracetamol and the other half will receive Ibuprofen.

DETAILED DESCRIPTION:
Paracetamol and Ibuprofen each relieve pain witf different mechanisms.

Paracetamol is termed a simple analgesic and an antipyretic. Despite enduring assertions that it acts by inhibition of cyclooxygenase (COX)-mediated production of prostaglandins, unlike non-steroidal anti-inflammatory drugs (NSAIDs).

Ibuprofen is the most commonly used and most frequently prescribed NSAID. It is a non-selective inhibitor of cyclo-oxygenase-1 (COX-1) and Cyclooxygenase-2 (COX-2).4 Although its anti inflammatory properties may be weaker than those of some other NSAIDs, it has a prominent analgesic and antipyretic role.

In our trial; The investigators aimed to compare intravenous Paracetamol and Ibuprofen in patient with Sciatica

* All patients eligible for the study(Approximately 200 patient with sciatica) were randomized to one of two groups:
* First Group: 1000 mg Paracetamol in 150 ml normal saline given as a slow intravenous infusion over 5 minutes.
* 100 ml of saline is removed before the addition of the 100 ml paracetamol to be the same volume.
* Second Group: 400 mg Ibuprofen in 150 ml normal saline given as a slow intravenous infusion over 5 minutes.
* Drug packs were prepared according to the computer-generated random number sequence to assign treatment allocations
* The allocation list was kept by the emergency nurse. Patients received the paracetamol or Ibuprofen medication schemes according to their random allocations.
* After enrollment and recording of baseline information, the next numbered study drug pack was obtained, and administered as a infusion over 5 minutes.
* Randomization was achieved by using computer software to generate random numbers.
* One researcher blinded to patient allocation observed the whole procedure and recorded the Sciatica pain scores.
* Patients in both groups received two types of medication in a similar manner (for example, 150 ml normal saline given as a slow intravenous infusion over 5 minutes), thus ensuring double blinding.
* Sciatica pain scores were recorded at 0, 15, and 30 min on a VAS of 1 to 10
* Rescue medication is given patients If the clinician think it's necessary within 30 minutes after study drug administration.
* All other medications required during the study also were recorded.

ELIGIBILITY:
Inclusion Criteria:

* Patients who presented with complaints of leg pain radiating the sciatic nerve tracings to the emergency services (Which may or may not be accompanied back pain),
* Positive Laseque test identified patients in physical examination,
* Patients whose complaints have started in the last week,
* Younger than 21 years old,
* Older than 65 years old.

Exclusion Criteria:

* Patients who have a leg or low back pain longer than a week Have a direct blunt trauma to the legs or lumbar area in the last week,
* Pretreatment linear 100-mm visual analog scale (VAS) pain score less than 40 mm,
* Patients who have drop foot, paralysis and other neurological symptoms in physical examination.
* Patients with blood pressure less than 90mmHg in the arrival of emergency services.
* Patients with malignancy, cauda equina syndrome, ankylosing spondylitis, rheumatoid arthritis or inflammatory arthritis contain any of the disease in his/her CV.
* Patients with any history of chronic pain syndrome.
* Patients who receive pain killers, antidepressants, anticonvulsants, muscle relaxants, steroids within 6 hours before the ED visit,
* Patients with a history of Substance Dependence or alcohol abuse
* Patients had a fever (>37.9)
* Allergy or previous adverse reaction to the studied drugs(Ibuprofen, Paracetamol), received agents to inhibit the secretion of acid (PPIs or histamine-2 receptor antagonists), antispasmodics, or nonsteroidal anti-inflammatory drugs
* were pregnant or breast-feeding,
* inability to comprehend the VAS evaluation,
* or refused to participate in the study

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2016-03; Primary Completion 2016-08 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
Reduction of Sciatica pain in Visual Analog Scale İn 30 minutes. | Sciatica pain scores will be recorded at 0, 15, and 30 min.
  this work tooks 6 mounts

SECONDARY OUTCOMES:
Adverse events | 30 minutes after the drug administered.
  30 minutes after the study drug administered

CONTACTS AND LOCATIONS:
Overall Officials: Mustafa SERINKEN, professor, Study Director — Pamukkale University; Cenker EKEN, associate professor, Study Director — Akdeniz University
Locations (1):
- Pamukkale University, Denizli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided